CLINICAL TRIAL: NCT05883644
Title: A Phase IIIb Single Arm, Open-label, Multicentre Study of Durvalumab and Tremelimumab as First Line Treatment in Participants With Advanced Hepatocellular Carcinoma (SIERRA)
Brief Title: Durvalumab and Tremelimumab as First Line Treatment in Participants With Advanced Hepatocellular Carcinoma (HCC)
Acronym: SIERRA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419CR00030; 2022-502012-37-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: liver cancer; human mAb; immunoglobulin G1 kappa subclass; STRIDE; Barcelona Clinic Liver Cancer (BCLC); Child-Pugh
MeSH Terms: conditions — Liver Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Phase IIIb Non-randomised and non-blinded single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab plus Tremelimumab (Experimental): Participants will receive a single priming dose of Tremelimumab plus Durvalumab at Day 1 (Week 0), followed by Durvalumab monotherapy starting at Week 4 and continuing until clinical progression, confirmed RECIST 1.1-defined radiological progression, unacceptable toxicity, withdrawal of consent, or any intervention discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Participants will receive 1500 mg at Day 1 and later receive as monotherapy starting at Week 4 for every 4 weeks through IV infusion
Drug: Tremelimumab — Participants will receive single dose of 300 mg through IV infusion at Day 1

SUMMARY:
This study will assess the safety and efficacy of Single Tremelimumab Regular Interval Durvalumab (STRIDE) as first-line therapy in participants with advanced unresectable HCC.

DETAILED DESCRIPTION:
This is a Phase IIIb, open-label, single arm, multicentre study to assess the safety and efficacy of STRIDE as first-line therapy in participants with advanced unresectable HCC who have one of the following:

1. Child-Pugh score B7 or B8 with a World Health Organisation Eastern Cooperative Oncology Group Performance Status (WHO/ECOG PS) of 0-1 at enrolment, or
2. Child-Pugh class A with a WHO/ECOG PS of 2 at enrolment, or
3. Child-Pugh class A with a WHO/ECOG PS of 0-1 and with evidence of chronic main trunk portal vein thrombosis at enrolment

Participants must not have received any prior systemic therapy for HCC. Participants may have previously received locoregional therapy (LRT) but must no longer be suitable for additional LRT. Any local treatment needs to have been completed at least 4 weeks prior to initiation of treatment. The study consists of 4 periods: screening (Day-28 to Day -1), Treatment period, safety follow-up and survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed unresectable HCC based on histopathological findings (prior histological verification confirming HCC is acceptable), or radiological findings in participants with cirrhosis where histopathological confirmation is not clinically feasible
* Must not have received prior systemic therapy for HCC
* Participants expected to live 12 weeks or more
* At least 1 measurable lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter with CT or MRI, and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines
* Must not be eligible for LRT for unresectable HCC.
* Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy LRT) or stage C
* Child-Pugh Score classification on liver disease and WHO/ECOG PS at enrolment complying one of the following:

  1. Child-Pugh score B7 or B8 with a WHO/ECOG PS of 0-1 at enrolment, without main trunk portal vein thrombosis.
  2. Child-Pugh class A with a WHO/ECOG PS of 2 at enrolment, without main trunk portal vein thrombosis (ie, ECOG PS 2 participants with main portal vein tumour thrombosis are excluded from this study).
  3. Child-Pugh class A with WHO/ECOG PS of 0-1 at enrolment and with chronic main trunk portal vein thrombosis
* Participants with hepatitis B virus (HBV) infection must be treated with antiviral therapy prior to enrolment.
* Participants with hepatitis C virus (HCV) infection must have confirmed diagnosis of HCV characterized by the presence of detectable HCV RNA or anti-HCV upon enrolment
* Adequate organ and bone marrow function
* Negative pregnancy test (serum) for women of childbearing potential.
* Female participants must be 1 year post-menopausal, surgically sterile, or using one highly effective form of birth control
* Male and Female participants and their partners must use an acceptable method of contraception.
* Body weight >30 kg

Exclusion Criteria:

* Any evidence of acute or uncontrolled diseases, chronic diverticulitis or previous complicated diverticulitis, or history of allogeneic organ transplant, which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol
* Refractory nausea and vomiting, chronic gastrointestinal (GI) disease, inability to swallow a formulated product, or previous significant bowel resection
* History of symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence, or
  2. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or lentigo maligna that has undergone potentially curative therapy, or
  3. Adequately treated carcinoma in situ without evidence of disease
* Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade > 1) caused by previous anticancer therapy
* Active or prior documented autoimmune or inflammatory disorders, autoimmune pneumonitis, and autoimmune myocarditis
* History of active primary immunodeficiency
* History of leptomeningeal carcinomatosis
* History of hepatic encephalopathy within the past 6 months or requirement for medications to prevent or control encephalopathy
* Active or prior documented GI bleeding (eg. esophageal varices or ulcer bleeding) within the past 6 months.
* Clinical judgement of acute main trunk portal vein thrombosis
* History of previous, or current, brain metastases or spinal cord compression
* Known fibrolamellar hepatocellular carcinoma (HCC), sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Clinically meaningful ascites
* Participants co-infected with HBV and HCV or co-infected with HBV and hepatitis D virus (HDV)
* Known to have tested positive for human immunodeficiency virus (HIV) or active tuberculosis infection
* Any concomitant medication known to be associated with Torsades de Pointes
* Prior exposure to immune-mediated therapy excluding therapeutic anticancer vaccines
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention" and "Major surgical procedure (as defined by the investigator) or significant traumatic injury within 4 weeks of the first dose of study intervention.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or 4 possibly related to treatment adverse events (PRAEs) | From the date of first dose of IMP until 6 months after the initiation of study intervention
  PRAE is defined as an AE which has been assessed by the investigator to be possibly related to IMP.
Objective response rate (ORR) | From the first dose of IMP until progression, or the last evaluable assessment in the absence of progression [approx. up to 33 months]
  ORR is defined as the number (%) of participants with a confirmed objective tumour response (complete response [CR] or partial response [PR]) as determined by the investigator per Response Evaluation Criteria in Solid Tumours, Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs), adverse event of special interest (AESIs), immune-mediated AEs (imAEs) | From screening until 90 days following discontinuation of the last dose of IMP [approx. up to 33 months]
  To assess the safety and tolerability of STRIDE in participants with advanced unresectable HCC
Overall Survival (OS) | From the date of the first dose of IMP until death [maximum follow-up approx. 33 months]
  OS is defined as the time from the date of the first dose of IMP until death due to any cause.
Progression-Free Survival (PFS) | From the date of the first dose of IMP until the date of objective PD or death [maximum follow-up approx. 33 months]
  PFS is defined as the time from the first dose of IMP until the date of objective PD (per RECIST 1.1 as assessed by the investigator) or death (by any cause in the absence of progression)
Disease Control Rate at Week 16 (DCR-16w) | At Week 16
  DCR-16w is defined as the percentage of participants who have a best objective response of complete response or partial response (by Week 16 + 7 days) or who have stable disease for at least 16 weeks (-7 days), following the start of study intervention as determined by the investigator per RECIST 1.1
Disease Control Rate at Week 24 (DCR-24w) | At Week 24
  DCR-24w is defined as the percentage of participants who have a best objective response of complete response or partial response (by Week 24 + 7 days) or who have stable disease for at least 24 weeks (-7 days), following the start of study intervention per RECIST 1.1
Duration of Response (DOR) | From the date of first documented response until the first date of documented progression or death in the absence of disease progression [approx. up to 33 months]
  DOR is defined as the time from the date of first documented response until the date of documented progression per RECIST 1.1, as assessed by the investigator or death in the absence of disease progression.
Duration of Treatment (DOT) | From the date of first dose of IMP to the date of last dose of IMP [approx. up to 33 months]
  DOT is defined as time on study intervention.
Time to deterioration in Health-Related Quality of Life (HRQoL), assessed using the EORTC QLQ C-30. | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Time to deterioration is defined as time from date of first dose of study intervention to the date of the first clinically meaningful deterioration (defined as a a decrease from baseline of at least 10 points for EORTC QLQ-C30 global HRQoL and functional scales, and an increase from baseline of at least 10 points for the EORTC QLQ-C30 symptom scales) that is confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration. The domains/scales of the EORTC QLQ-C30 prioritized include global health status/QoL, functioning (physical), multi-term symptom (fatigue) and single item symptoms (appetite loss and nausea). Final scores range from 0 to 100, where higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Clinically meaningful change from baseline in HRQoL as assessed by EORTC QLQ C-30 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Clinically meaningful change from baseline in global health status/QoL, symptoms and function score (categorized as improvement, no change or deterioration) is defined as an absolute change in the score from baseline of ≥ 10 for scales from the EORTC QLQ-C30 to assess disease and treatment related symptoms and HRQoL.The domains/scales of the EORTC QLQ-C30 prioritized include global health status/QoL, functioning (physical), multi-term symptom (fatigue) and single item symptoms (appetite loss and nausea). Final scores range from 0 to 100, where higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Best overall response for HRQoL as assessed by EORTC QLQ C-30 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Best overall response for global health status/QoL, function and symptom (fatigue) will be derived as the best response the participant achieved, based on evaluable electronic patient-reported outcome (ePRO) data collected during the study period to assess disease and treatment related symptoms and HRQoL. The domains/scales of the EORTC QLQ-C30 prioritized include global health status/QoL, functioning(physical), multi-term symptom (fatigue) and single item symptoms (appetite loss and nausea). Final scores range from 0 to 100, where higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Change from baseline in HRQoL as assessed by EORTC QLQ C-30 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Change from baseline of global health status/QoL, symptom and functioning scores to assess disease and treatment related symptoms and HRQoL. The domains/scales of the EORTC QLQ-C30 prioritized include global health status/QoL, functioning(physical), multi-term symptom (fatigue) and single item symptoms(appetite loss and nausea). Final scores range from 0 to 100, where higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Time to deterioration in HRQoL as assessed by EORTC QLQ-HCC18 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Time to deterioration is defined as time from date of first dose of study intervention to the date of the first clinically meaningful deterioration (defined as an increase from baseline of at least 10 points for EORTC QLQ-HCC18) that is confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration. The QLQ-HCC18 is an HCC-specific module from the EORTC comprising 18 questions to assess HCC symptoms. The module includes 6 multi-item domain scales and 2 single-item scales. Final scores range from 0 to 100 where higher scores indicate a greater level of symptom severity and a poorer HRQoL. The items prioritized are single items shoulder pain, abdominal pain and abdominal swelling.
Clinically meaningful change from baseline in HRQoL as assessed by EORTC QLQ-HCC18 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Clinically meaningful change from baseline (categorized as improvement, no change or deterioration) is defined as an absolute change in the score from baseline of ≥ 10 for scales/items from QLQ-HCC18 to assess disease-related symptoms. The single items prioritized are shoulder pain, abdominal pain and abdominal swelling. The EORTC QLQ-HCC18 module is an 18-item questionnaire. All questions have a 4-point scale: "Not at all," "A little," "Quite a bit," and "Very much." For each of the 8 domains (6 multiple-item scales and 2 single-item scales), final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms and worse symptom or a poorer HRQoL.
Best overall response for HRQoL as assessed by EORTC QLQ-HCC18 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Best overall response in single-item symptoms (shoulder pain, abdominal pain, abdominal swelling) will be derived as the best response the participant achieved, based on evaluable ePRO data collected during the study period to assess disease-related symptoms. The single items prioritized are shoulder pain, abdominal pain and abdominal swelling. The EORTC QLQ-HCC18 module is an 18-item questionnaire. All questions have a 4-point scale: "Not at all," "A little," "Quite a bit," and "Very much." For each of the 8 domains (6 multiple-item scales and 2 single-item scales), final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms and worse symptom or a poorer HRQoL.
Change from baseline in HRQoL as assessed by EORTC QLQ-HCC18 | Every 8 weeks from date of first dose of IMP for the first 48 weeks and then every 12 weeks thereafter until treatment discontinuation and 90 days after last dose during safety follow-up [approx. up to 33 months]
  Change from baseline assessment in EORTC QLQ-HCC18 scale/item score at each post baseline assessment. The prioritized single items scores are shoulder pain, abdominal pain and abdominal swelling. The EORTC QLQ-HCC18 module is an 18-item questionnaire. All questions have a 4-point scale: "Not at all," "A little," "Quite a bit," and "Very much." For each of the 8 domains (6 multiple-item scales and 2 single-item scales), final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms and worse symptom or a poorer HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chan, MD, Principal Investigator — Department of Clinical Oncology, Chinese University of Hong Kong; Lorenza Rimassa, MD, Principal Investigator — Humanitas Cancer Centre, IRCCS Humanitas Research Hospital
Locations (35):
- United States (3):
  - Research Site, La Jolla, California
  - Research Site, Shreveport, Louisiana
  - Research Site, Detroit, Michigan
- France (5):
  - Research Site, Bobigny
  - Research Site, Clichy
  - Research Site, Créteil
  - Research Site, Marseille
  - Research Site, Rennes
- Germany (4):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Frankfurt
  - Research Site, Lübeck
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Italy (6):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Rozzano
  - Research Site, Turin
- Japan (6):
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Matsuyama
  - Research Site, Musashino-shi
  - Research Site, Osakasayama-shi
  - Research Site, Yokohama
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Gyeonggi-do
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Pamplona
- Research Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home